CLINICAL TRIAL: NCT06657924
Title: Preoperative Tranexamic Acid (TXA) to Prevent Bleeding in Patients Undergoing Major Colorectal Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kristen Ban (Other)
Responsible Party: Sponsor-Investigator, Kristen Ban, Assistant Professor of Surgery, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB 24-896
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Bleeding; Colorectal Disorders; Thromboembolism; Tranexamic Acid
Keywords: Tranexamic Acid; TXA; Bleeding; Colorectal Surgery; Thromboembolism
MeSH Terms: conditions — Hemorrhage; Thromboembolism | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Intervention (TXA) and control (no TXA) cohorts
Masking Description: Pragmatic (non-blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid (Experimental): TXA administered as a 1 gram IV bolus in 100ml of normal saline administered over 10 minutes at the start and end of the surgery for a total of 2 grams TXA
  Interventions: Drug: Tranexamic acid
- Control (no tranexamic acid) (No Intervention): Standard of care

INTERVENTIONS:
Drug: Tranexamic acid — 1 gram IV bolus in 100ml of normal saline administered over 10 minutes at the start and end of the surgery for a total of 2 grams TXA
  Arms: Tranexamic Acid

SUMMARY:
The goal of this prospective pragmatic randomized clinical trial is to determine if preoperative administration of tranexamic acid (TXA) reduces bleeding during and after major colorectal surgery. The primary questions are:

* Does TXA reduce bleeding during and after surgery (change in hemoglobin from before surgery to lowest value after surgery within 30 days)
* Does TXA reduce bleeding complications within 30 days of surgery (blood transfusion, return to the operating room or procedural intervention for bleeding, death due to bleeding)
* Does TXA increase the risk of thromboembolic complications within 30 days of surgery (cerebrovascular accident, myocardial infarction, deep venous thrombosis, pulmonary embolism)

Researchers will compare preoperative TXA to no TXA to answer the above questions.

Participants who receive TXA will receive 1 g TXA IV at the beginning and end of surgery in the operating room.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 18 years or older
2. Undergoing elective or non-elective inpatient abdominal and pelvic colorectal surgery

Exclusion Criteria:

1. Creatinine clearance less than 30 mL/minute
2. Long-term dialysis
3. Known defective color vision (color blind)
4. Pregnancy
5. History of venous or arterial thromboembolism, or active thromboembolic disease
6. Disseminated intravascular coagulation (DIC) - clinically suspected and/or confirmed by platelet count on CBC, fibrinogen, INR and PTT.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 394 (Estimated)
Dates: Start 2025-02-11 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative change in hemoglobin | 60 days
  Preoperative to lowest postoperative within 30 days of surgery

SECONDARY OUTCOMES:
Rate of composite bleeding complication | Within 30 days postop
  Bleeding requiring transfusion, bleeding prompting medication to be held for DVT prophylaxis or therapeutic anticoagulation, bleeding requiring return to the operating room or procedural intervention, mortality secondary to bleeding
Rate of composite thromboembolic event | Within 30 days postop
  Thromboembolic cerebrovascular accident (CVA), myocardial infarction (MI), deep venous thrombosis (DVT), pulmonary embolism (PE)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen A Ban, MD MS, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Fairview Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No